CLINICAL TRIAL: NCT03237117
Title: Effect of Growth Hormone on Uterine Receptivity in Women With RIF in an Oocyte Donation Program: a Randomized Controlled Trial
Brief Title: Effect of Growth Hormone on Uterine Receptivity in Women With RIF in an Oocyte Donation Program
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Competence Centre on Health Technologies (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Signe Altmäe, Senior researcher, Competence Centre on Health Technologies
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MarGen
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: 105 infertile women are enrolled in the randomized controlled trial: 70 women are with a history of RIF with donated oocytes and 35 infertile women undergoe the first oocyte donation attempt. 35 RIF patients are treated with GH (GH patients, study group) while the rest 35 RIF patients (non-GH patients, negative control group) and 35 first-attempt patients (positive control group) are not.
Who Masked: Participant, Care Provider
Masking Description: The assignments are concealed in sealed opaque envelopes until the time of enrollment: group I (GH patients) and group II (non-GH patients). All injections are performed by an independent nurse who is informed by the trial coordinator of each woman´s number and the treatment allocation. Consequently, both the clinician and the patients are blinded as to the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GH group (Experimental): 35 women with a history of RIF with donated oocytes. For receiving donated oocytes, the women are treated with progressively increasing doses of oral estradiol followed by intravaginal progesterone after previous pituitary desensitization with GnRH agonist. Additionally, these patients are co-treated with growth hormone (GH).
  Interventions: Biological: Growth Hormone (GH)
- non-GH group (Active Comparator): 35 women with a history of RIF with donated oocytes. For receiving donated oocytes, the women are treated with progressively increasing doses of oral estradiol followed by intravaginal progesterone after previous pituitary desensitization with GnRH agonist. The treatment protocol is identical to the GH group, only that no GH is added.
  Interventions: Biological: Growth Hormone (GH)
- positive control group (No Intervention): 35 infertile women undergoing their first oocyte donation attempt are included as a positive control group. Women receiving donated oocytes are treated with progressively increasing doses of oral estradiol followed by intravaginal progesterone after previous pituitary desensitization with GnRH agonist. The treatment protocol is identical to the non-GH group, with no GH added.

INTERVENTIONS:
Biological: Growth Hormone (GH) — to evaluate the effect of GH administration in the donated oocyte recipient program among women with RIF (repeated implantation failure)
  Arms: GH group; non-GH group

SUMMARY:
105 infertile women are enrolled in the randomized controlled trial: 70 women with a history of RIF with donated oocytes and 35 infertile women undergoing the first oocyte donation attempt. Women receiving donated oocytes are treated with progressively increasing doses of oral estradiol followed by intravaginal progesterone after previous pituitary desensitization with GnRH agonist. 35 RIF patients are treated with GH (GH patients) while the rest 35 RIF patients (non-GH patients) and 35 first-attempt patients (positive control group) are not.

DETAILED DESCRIPTION:
This study includes in total 105 infertile couples treated by assisted reproduction with oocyte donation. Seventy couples that have experienced at least two previous failures with this approach at our clinic are referred to as recurrent implantation failure (RIF) patients throughout this study. Thirty five of these couples are included in the GH-treatment protocol, while the remaining 35 couples are treated in a usual way (non-GH group). Other 35 couples, treated in the same period and undergoing their first oocyte donation attempt, are included as a positive control group.

RIF patients are randomly allocated into two groups (labeled I and II). Then the assignments are concealed in sealed opaque envelopes until the time of enrollment: group I (GH patients) and group II (non-GH patients). All injections are performed by an independent nurse who is informed by the trial coordinator of each woman´s number and the treatment allocation. Consequently, both the clinician and the patients are blinded as to the treatment received. The positive control (non-RIF) group is created by allocating all consecutive couples undergoing their first oocyte donation attempt. This allocation started immediately after the allocation of the first RIF couple and will be terminated as soon as 35 cases are enrolled.

Ovarian stimulation of the oocyte donors is as follows: oocyte donors are stimulated with the use of a long GnRH agonist protocol and human recombinant FSH (Puregon or Gonal F). Human menopausal gonadotropin (Menopur) is added when blood LH concentration, which is repeatedly determined during ovarian stimulation, falls below 1 IU/l. Final oocyte maturation is triggered by subcutaneous injection of 250 micrograms recombinant hCG (Ovitrelle), when at least 5 follicles measure 18 mm or more. Ovarian puncture for oocyte recovery is performed 36.5 h after recombinant hCG injection.

Oocyte recipients are treated with progressively increasing doses of orally administered pure estradiol (Provames) or estradiol valerate (Progynova) after previous pituitary desensitization with a single injection of the long-acting preparation of GnRH agonist triptorelin (Decapeptyl 3,75 mg). The interval between triptorelin injection and the beginning of oral estradiol treatment is ranging between 8 and 20 days. This interval is determined individually, in each case, in view of the optimal synchronization of the recipient's endometrial development and the follicular growth of the corresponding donor.

ELIGIBILITY:
Inclusion Criteria for oocyte recipients:

* age below 51 years
* 2 or more previous implantation failures in oocyte donation program
* voluntary participation

Inclusion Criteria for oocyte donors:

* age up to 25 year
* healthy
* voluntary participation

Exclusion Criteria:

* cancellation of the treatment
* no wish to participate any longer

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 2010-2017
  Pregnancy rate is calculated as the number of patients with positive beta-hCG test divided by the number of patients in whom embryos were transferred
live birth rate | 2010-2017
  Live birth rate is calculated as the number of babies born by the number of embryos transferred
live delivery rate | 2010-2017
  live delivery rate is obtained by dividing the number of births with the number of transfers

SECONDARY OUTCOMES:
ongoing pregnancy rate | 2010-2017
  ongoing pregnancy rate is the number of patients with the presence of fetal heart activity divided by the number of transfer procedures
implantation rate | 2010-2017
  Implantation rate is the number of embryonic sacs detected on ultrasound divided by the number of embryos transferred
ongoing implantation rate | 2010-2017
  ongoing implantation rate is calculated by dividing the number of living fetuses developing beyond 20 weeks divided by the number of embryos transferred
miscarriage rate | 2010-2017
  miscarriage rate is defined as the number of miscarriages before 20 weeks divided by the number of women with a positive pregnancy test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No
No other IPD is foreseen than scientific publications.